CLINICAL TRIAL: NCT02275260
Title: Reduction of AF Ablation Induced Thrombo-Embolic Incidence Pilot Study (REDUCE-TE Pilot)
Brief Title: Reduction of AF Ablation Induced Thrombo-Embolic Incidence Pilot Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The required number of endpoints will be obtained with a sample size lower than initially planned.
Sponsor: Biotronik SE & Co. KG (Industry)
Collaborators: University Hospital Heidelberg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: EP025
Record Dates: First submitted 2014-10-21; First posted 2014-10-27 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2018-05

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Echocardiography, Transesophageal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All patients (Experimental): All patients undergo cerebral Diffusion-Weighted Magnetic Resonance Imaging (DW-MRI), Transesophageal (or Intracardial) Echocardiography and paperbased neurocognitive testing
  Interventions: Device: Cerebral Diffusion-Weighted Magnetic Resonance Imaging; Device: Transesophageal Echocardiography; Other: Paperbased neurocognitive testing

INTERVENTIONS:
Device: Cerebral Diffusion-Weighted Magnetic Resonance Imaging — Patients undergo a cerebral Diffusion-Weighted Magnetic Resonance Imaging (DW-MRI)
  Other Names: 1.5-3 T machine capable of Diffusion-Weighted MRI
Device: Transesophageal Echocardiography — Patients undergo a Transesophageal Echocardiography prior to the ablation itself
  Other Names: Any Transesophageal Echocardiography machine
Other: Paperbased neurocognitive testing — To assess the impact of PVI on the patient's neurocognitive status
  Other Names: STATE questionnaire, d2 test, visual VVM2, MOCA subtest

SUMMARY:
The REDUCE-TE Pilot study is an international, multicenter, prospective, single arm study to compare the AlCath Flux eXtra Gold ablation catheter regarding the prevention of new subclinical cerebral thromboembolic lesions after Pulmonary Vein Isolation to historical data from the literature.

ELIGIBILITY:
Inclusion Criteria:

* Electrocardiographically documented, symptomatic paroxysmal AF.
* Patients with indication for left atrial ablation of AF according to ESC guidelines for the management of atrial fibrillation.
* Anticoagulation according to clinical routine using coumarin derivates with target INR between 2.0 and 3.0 at least 3 weeks prior to the scheduled ablation procedure or novel oral anticoagulants (NOACs).
* Geographically stable for the duration of the study.
* Willingness and ability to perform written informed consent

Exclusion Criteria:

* Long standing persistent or persistent AF
* CHA2DS2-VASc score ≥ 5
* Prior ischemic stroke or Transient Ischemic Attack
* Previous Pulmonary Vein ablation
* Contraindication for anticoagulation therapy
* Contraindication for Diffusion-Weighted MRI
* Claustrophobia
* Contraindication for transesophageal echocardiography (TEE) or intracardiac echocardiography (ICE, if TEE not possible)
* Implanted cardiovascular device, including but not limited to an atrial or ventricular pacemaker or defibrillator leads, artificial valves, stents, septal or LAA occluders
* Acute coronary syndrome < 3 months prior to scheduled ablation
* Moderate to severe valvular heart disease
* LA size > 55 mm (confirming echo at maximum 3 months old)
* Patients with non-controlled heart failure or patients with current and recent (< 1 month prior to ablation) heart failure
* Ejection fraction < 35% (confirming echo at maximum 3 months old)
* Conditions that prevent patient's participation in neurocognitive assessment (at physician's discretion)
* Female patients who are pregnant or breast feeding or plan a pregnancy during the course of the study
* Any limitation to contractual capability
* Simultaneous participation in another study
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-02-08 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Thromboembolic lesions | 1-3 days
  The occurrence of one or more new subclinical cerebral thromboembolic lesions after Pulmonary Vein Isolation assessed by Diffusion-Weighted MRI

SECONDARY OUTCOMES:
Neurocognitive status | Baseline, 1-3 days and 3 months
  To assess the impact of PVI on the patient's neurocognitive status measured by a testing battery including the STATE questionnaire, d2 test of attention, visual part of the visual and verbal memory test (VVM2) and Montreal Cognitive Assessment (MOCA) subtest
Peri-procedural serious adverse events | Within 24 hours after ablation
  Any serious adverse event occurring during the ablation procedure and within 24 hours from completion of the procedure
Post-procedural clinical TE events | 3 months period
  Composite endpoint: Occurrence of Transient Ischemic Attack and/or Ischemic Stroke and/or Systemic Embolism during the three months post-ablation period (excluding peri-procedural events)

OTHER OUTCOMES:
Acute procedural success rate | During ablation
  Acute procedural success of Pulmonary Vein Isolation, defined as electrical isolation of all Pulmonary Veins (entrance block)
Success of Pulmonary Vein Isolation | 3 months
  Three months ablation success, defined as freedom from symptomatic AF recurrences off antiarrhythmic drug therapy assessed to three-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Dipen Shah, Prof. Dr., Study Chair — Hôpitaux Universitaires de Genève, Switzerland; Boris Schmidt, PD Dr., Study Chair — Cardioangiologisches Centrum Bethanien, Germany
Locations (14):
- Czechia (2):
  - Ceske Budejovice Hospital, České Budějovice
  - Institute for Clinical and Experimental Medicine (IKEM), Prague
- Germany (8):
  - Kerckhoff-Klinik, Bad Nauheim
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - Charité Campus Benjamin Franklin, Berlin
  - Charité Campus Virchow, Berlin
  - Cardioangologisches Centrum Bethanien (CCB), Frankfurt am Main
  - Universität Leipzig, Leipzig
  - Deutsches Herzzentrum München des Freistaates Bayern, Munich
  - Peter Osypka Herzzentrum München, Munich
- Semmelweis Medical University, Budapest, Hungary
- Netherlands (2):
  - OLVG - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Haga Ziekenhuis, The Hague
- Hôpitaux Universitaires de Genève, Geneva, Switzerland

REFERENCES:
- [Background] Akca F, Zima E, Vegh EM, Szeplaki G, Skopal J, Hubay M, Lendvai Z, Merkely B, Szili-Torok T. Radiofrequency ablation at low irrigation flow rates using a novel 12-hole gold open-irrigation catheter. Pacing Clin Electrophysiol. 2013 Nov;36(11):1373-81. doi: 10.1111/pace.12215. Epub 2013 Jul 22. PMID 23875670
- [Background] Balazs T, Laczko R, Bognar E, Akman S, Nagy P, Zima E, Dobranszky J, Szili-Torok T. Ablation time efficiency and lesion volume - in vitro comparison of 4 mm, non irrigated, gold- and platinum-iridium-tip radiofrequency ablation catheters. J Interv Card Electrophysiol. 2013 Jan;36(1):13-8; discussion 18. doi: 10.1007/s10840-012-9743-9. Epub 2012 Oct 26. PMID 23100094
- [Background] Linhart M, Liberman I, Schrickel JW, Mittmann-Braun EL, Andrie R, Stockigt F, Kreuz J, Nickenig G, Lickfett LM. Superiority of gold versus platinum irrigated tip catheter ablation of the pulmonary veins and the cavotricuspid isthmus: a randomized study comparing tip temperatures and cooling flow requirements. J Cardiovasc Electrophysiol. 2012 Jul;23(7):717-21. doi: 10.1111/j.1540-8167.2011.02267.x. Epub 2012 Mar 19. PMID 22429859
- [Background] Lewalter T, Weiss C, Spencker S, Jung W, Haverkamp W, Willems S, Deneke T, Kautzner J, Wiedemann M, Siebels J, Pitschner HF, Hoffmann E, Hindricks G, Zabel M, Vester E, Schwacke H, Mittmann-Braun E, Lickfett L, Hoffmeister S, Proff J, Mewis C, Bauer W; AURUM 8 Study Investigators. Gold vs. platinum-iridium tip catheter for cavotricuspid isthmus ablation: the AURUM 8 study. Europace. 2011 Jan;13(1):102-8. doi: 10.1093/europace/euq339. Epub 2010 Sep 28. PMID 20876601